CLINICAL TRIAL: NCT07139860
Title: Artificial Intelligence System for Early Warning of Adverse Events in Acute Myocardial Infarction
Acronym: AIEWAEAMI
Status: Recruiting | Type: Observational
Sponsor: Hui Chen (Other)
Responsible Party: Sponsor-Investigator, Hui Chen, PHD, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: BFH2023063001
Record Dates: First submitted 2025-08-22; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Acute Myocardial Infarction With ST Elevation; Intelligent Management Platform; Early Warning
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BFH: group1
- AZH: group2

SUMMARY:
The goal of this observational study is to learn about the effectiveness of an artificial intelligence-based early warning system for predicting adverse events in patients with acute myocardial infarction (AMI). The main question it aims to answer is:

Does an AI-based early warning system improve the assessment and prediction of adverse events across the full course of AMI care (from prevention to diagnosis, treatment, and rehabilitation)?

Participants who are receiving routine medical care for AMI in tertiary hospitals will have their multimodal medical data (clinical records, diagnostic tests, imaging, treatment pathways) collected and analyzed. Data will be integrated using innovative cross-modal representation methods and predictive models. The study will follow patients during their hospital stay and subsequent clinical follow-up to evaluate the feasibility, accuracy, and clinical value of the AI-based early warning system.

ELIGIBILITY:
Inclusion Criteria:

* 1. Hospitalized patients who meet the diagnostic criteria for acute myocardial infarction. 2. Patients who agree to participate and sign the informed consent form.

Exclusion Criteria:

* 1. Patients with terminal malignant tumors and an expected survival time of less than 3 months. 2. Patients with complete disability and inability to communicate. 3. Patients unable to comply with follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Retrospective Study Population:
     Data were obtained from the Cardiovascular Center Database (CBDBank) of Beijing Friendship Hospital. CBDBank is a continuously collected sample dataset of patients with acute coronary syndrome since January 2013. A total of 1,000 patients with acute myocardial infarction admitted to Beijing Friendship Hospital, Capital Medical University, from January 2017 to December 2019 were included in the retrospective cohort. After discharge, all patients received scheduled telephone follow-ups at 1 month, 3 months, 6 months, and annually thereafter, with continuous follow-up for 3 years.
  2. Prospective Study Population:
  A total of 800 patients with acute myocardial infarction admitted to the Cardiovascular Center of Beijing Friendship Hospital from July 2023 to July 2026 will be enrolled in the prospective cohort. Randomization will be performed using random codes, and prognosis prediction will be conducted using either the predictive system or traditional met
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MACCE | 1-3 years
  Cardiac death
  All-cause mortality
  Malignant arrhythmia
  Non-fatal recurrent myocardial infarction
  Non-fatal stroke
  Unplanned repeat revascularization
  Rehospitalization for heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China